CLINICAL TRIAL: NCT06459232
Title: Baseline Characteristics, Adherence, and Persistence Among Multiple Sclerosis Patients Treated With FDA-approved Disease-Modifying Therapies
Brief Title: Characteristics, Adherence, and Persistence Among Multiple Sclerosis Patients Treated With Disease-Modifying Therapies
Status: Completed | Type: Observational
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: CBAF312AUS16
Record Dates: First submitted 2024-06-10; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Multiple Sclerosis (MS) Cohort: Adult MS patients with at least 1 claim of siponimod or an MS-related FDA-approved DMT.

SUMMARY:
This retrospective, observational cohort study used administrative claims data contained in the International Business Machines (IBM)® Truven Marketscan® Research Databases to describe demographic, clinical, and treatment characteristics in patients with multiple sclerosis (MS) who were initiated on siponimod, and other Food and Drug Administration (FDA)-approved disease-modifying therapies (DMTs). The study time period was from March 2018 through June 2020 (most recent available data) and included a 1-year baseline period and a variable-length follow-up period (a minimum of 6 months follow-up required for post-index outcomes). The index date was defined as the date of the first claim for siponimod or other MS-specific treatment on or after March 2019.

The data analysis was performed on a combination of early view and standard view data. The initial data analysis was from Standard Marketscan data used for patients with index data prior to the year 2019. Both standard view and early view data were used for patients indexed after January 1, 2019. The early view data provided additional visibility as it contains an additional 2 quarters of data compared to standard data.

ELIGIBILITY:
Inclusion criteria

* With 1 or more claims of siponimod or MS-related FDA-approved DMT during the index calendar year. The date of first claim was the index date.
* With 1 or more MS diagnosis for 12 months prior to the index date [inclusive].
* Were continuously enrolled in pharmacy and medical benefits for 12 months prior to the index date [inclusive].
* Include patients who were 18 years or older on the index date.
* Include patients continuously enrolled in pharmacy and medical benefits from the index date [inclusive] to 6 months/12 months post-index date.

Exclusion criteria

• Patients with 1 or more claims of index drug within 12 months prior to index date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Number of Patients with a Minimum of 6 Months Follow-up by Disease-Modifying Therapy (DMT) Use | Baseline, defined as the 12 months prior to the first observed MS therapy claim (index date)
Number of Patients with a Minimum of 12 Months Follow-up by DMT Use | Baseline, defined as the 12 months prior to the first observed MS therapy claim (index date)

SECONDARY OUTCOMES:
Mean Age | Index date, defined as the date of the first claim for siponimod or MS-specific therapy
Number of Patients with a Minimum of 6 Months Follow-up by Age Group | Index date, defined as the date of the first claim for siponimod or MS-specific therapy
  Age group categories included:
  * 18-34 years
  * 35-44 years
  * 45-54 years
  * 55-64 years
  * 65+ years
Number of Patients with a Minimum of 12 Months Follow-up by Age Group | Index date, defined as the date of the first claim for siponimod or MS-specific therapy
  Age group categories included:
  * 18-34 years
  * 35-44 years
  * 45-54 years
  * 55-64 years
  * 65+ years
Number of Patients with a Minimum of 6 months Follow-up by Gender | Index date, defined as the date of the first claim for siponimod or MS-specific therapy
Number of Patients with a Minimum of 12 months Follow-up by Gender | Index date, defined as the date of the first claim for siponimod or MS-specific therapy
Number of Patients with a Minimum of 6 Months Follow-up by Geographical Region | Index date, defined as the date of the first claim for siponimod or MS-specific therapy
Number of Patients with a Minimum of 12 Months Follow-up by Geographical Region | Index date, defined as the date of the first claim for siponimod or MS-specific therapy
Number of Patients with a Minimum of 6 Months Follow-up by Insurance Plan Type | Index date, defined as the date of the first claim for siponimod or MS-specific therapy
Number of Patients with a Minimum of 12 Months Follow-up by Insurance Plan Type | Index date, defined as the date of the first claim for siponimod or MS-specific therapy
Number of Patients with a Minimum of 6 Months Follow-up by Health Plan Type | Index date, defined as the date of the first claim for siponimod or MS-specific therapy
Number of Patients with a Minimum of 12 Months Follow-up by Health Plan Type | Index date, defined as the date of the first claim for siponimod or MS-specific therapy
Percentage of Patients with MS Relapses | Baseline, defined as the 12 months prior to the first observed MS therapy claim
Mean Charlson Comorbidity Index (CCI) Score | Baseline, defined as the 12 months prior to the first observed MS therapy claim
  CCI predicts the ten-year mortality for a patient who may have a range of comorbid conditions. Comorbidity was assessed using the CCI, categorized as low (0-1) and high (≥2).
Percentage of Patients with a Minimum of 6 Months Follow-up by Disability Level | Baseline, defined as the 12 months prior to the first observed MS therapy claim
  Disability levels included: No symptoms, Mild, Moderate, and Severe.
Percentage of Patients with a Minimum of 12 Months Follow-up by Disability Level | Baseline, defined as the 12 months prior to the first observed MS therapy claim
  Disability levels included: No symptoms, Mild, Moderate, and Severe.
Percentage of Patients with a Minimum of 6 Months Follow-up by Most Observed Comorbidities | Baseline, defined as the 12 months prior to the first observed MS therapy claim
Percentage of Patients with a Minimum of 12 Months Follow-up by Most Observed Comorbidities | Baseline, defined as the 12 months prior to the first observed MS therapy claim
Number of Patients with a Minimum of 6 Months Follow-up by Type of Prior Disease-Modifying Therapy (DMT) | Baseline, defined as the 12 months prior to the first observed MS therapy claim
Number of Patients with a Minimum of 12 Months Follow-up by Type of Prior DMT | Baseline, defined as the 12 months prior to the first observed MS therapy claim
Mean Proportion of Days Covered (Adherence) for Patients with a Minimum of 6 Months Follow-up | 6 months post-index date (defined as date of the first claim for siponimod or other MS-specific treatment)
  Proportion of days covered was calculated as the number of days in the follow-up period that the patient had index medication on hand, divided by the total number of days in the follow-up period.
Mean Proportion of Days Covered (Adherence) for Patients with a Minimum of 12 Months Follow-up | 12 months post-index date (defined as date of the first claim for siponimod or other MS-specific treatment)
  Proportion of days covered was calculated as the number of days in the follow-up period that the patient had index medication on hand, divided by the total number of days in the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States